CLINICAL TRIAL: NCT00686491
Title: Center of Excellence in CardioRespiratory Health of High-level Athletes: Evaluation of Long-term Effects of Training.
Brief Title: Respiratory Health of Elite Athletes
Acronym: cold air
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Dr Louis-Philippe BOULET, Institut universitaire de cardiologie et de pneumologie de Québec
Other Study IDs: CER 20141
Record Dates: First submitted 2008-05-26; First posted 2008-05-29 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Asthma; Cardiovascular Diseases; Metabolic Diseases
Keywords: Asthma; Environment; Type of sport; Cardiovascular disease; Athletes
MeSH Terms: conditions — Asthma; Cardiovascular Diseases; Metabolic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum - plasma - sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1: Triathletes
- 2: Cold air athletes
- 3: Swimmers
- 4: Other sports elite athletes
- 5: Control subjects

SUMMARY:
Eleven National Sports Teams are located in the Quebec Metropolitan Area. In these groups, many athletes are aiming for Olympic medals in Beijing 2008 and Vancouver 2010 Olympic Games. A consultation of the coaches of these National Teams revealed that although a large proportion of these athletes present various cardio-respiratory symptoms, they do not have a rapid access to a systematic medical evaluation and follow-up. Furthermore, little is done in regard to prevention and optimization of treatment of pulmonary and cardiac conditions in the elite athlete's population of the Quebec area.

Cardiorespiratory problems are therefore commonly found in high-level athletes. However, these pathologies are not well characterized in athletes and the associated symptoms often not well perceived. These problems can be serious and it is important to detect them before they appear1 while setting up a systematic medical follow-up. Health professionals should monitor health of the young athletes and help to reduce the risks associated with high level exercise. The following project is an evaluation and follow-up program of high-level athletes, aiming at gathering key-information on long-term effects of high-level training on cardio-respiratory and metabolic parameters. Our aims will be

1. to establish a long-term program of systematic evaluation and follow-up of cardiorespiratory health and performance of high elite athletes.
2. to evaluate the prevalence of respiratory, circulatory and metabolic problems among high-level athletes
3. to evaluate the effects of treatments on cardiorespiratory conditions and exercise performance in athletes who need asthma medication.

ELIGIBILITY:
Inclusion Criteria:

* Athletes training more than 10 hours per week-

Exclusion Criteria:

* asthma or other pathologies that may interfere with the study
* Smokers
* Obese of with a BMI more than 29

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Athletes training in the province of Quebec. Controls from Quebec schools and universities.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2007-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul POIRIER, MD, Principal Investigator — Hôpital LAval
Locations (1):
- Centre de recherche de l'Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada

REFERENCES:
- [Derived] Bougault V, Blouin E, Turmel J, Boulet LP. Airway response to methacholine following eucapnic voluntary hyperpnea in athletes. PLoS One. 2015 Mar 19;10(3):e0121781. doi: 10.1371/journal.pone.0121781. eCollection 2015. PMID 25789614
- [Derived] Turmel J, Bougault V, Boulet LP, Poirier P. Exaggerated blood pressure response to exercise in athletes: dysmetabolism or altered autonomic nervous system modulation? Blood Press Monit. 2012 Oct;17(5):184-92. doi: 10.1097/MBP.0b013e3283573509. PMID 22828668
- [Derived] Bougault V, Turmel J, Boulet LP. Bronchial challenges and respiratory symptoms in elite swimmers and winter sport athletes: Airway hyperresponsiveness in asthma: its measurement and clinical significance. Chest. 2010 Aug;138(2 Suppl):31S-37S. doi: 10.1378/chest.09-1689. Epub 2010 Apr 2. PMID 20363843